CLINICAL TRIAL: NCT07157839
Title: Detection of Elevated Plasma pTau217 in Donated Human Blood Samples: Implications for Blood Transfusion Safety
Brief Title: Phosphorylated Tau Levels in Donated Blood
Acronym: pTIDB
Status: Recruiting | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Zhongcong Xie, Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-25-0343; 5R01AG062509 (NIH)
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Alzheimer&Amp;#39;s Disease
Keywords: Phosphorylated Tau, donated blood, Alzheimer's disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Donated plasma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Alzheimer's disease (AD) is characterized by the accumulation of tau pathology, and blood-based biomarkers such as phosphorylated tau-217 (pTau217) have been identified as sensitive and specific predictors of AD risk. Recent studies suggest that individuals with elevated pTau217 levels may be at increased risk for developing AD and cognitive dysfunction. This observational study will examine donated human plasma samples to determine whether some units of donated blood contain abnormally elevated pTau217 concentrations. The overarching goal is to evaluate whether transfusion of blood with higher pTau217 may pose risks to recipients and whether such units should be avoided in clinical use.

DETAILED DESCRIPTION:
Study Type:

Observational (Laboratory-based biomarker study; no human intervention)

Study Design:

* Model: Cross-sectional
* Time Perspective: Prospective
* Sample Source: Donated human blood plasma samples obtained through a blood bank
* Enrollment: ~250 plasma samples; ~20 plasma samples of AD patients and ~20 plasma samples of normal control participants, where are purchased from BioIVT (Westbury, NY, USA).

Official Title:

Observational Measurement of pTau217 in Donated Human Plasma Samples

Primary Objective:

To determine the prevalence of elevated plasma pTau217 levels in donated blood.

Secondary Objectives:

1. To compare pTau217 concentrations with total Tau to assess biomarker distribution in donated blood.
2. To generate preliminary data on whether pTau217 screening could be relevant to transfusion safety guidelines.

Primary Outcome Measure:

* Proportion of blood samples with plasma pTau217 levels exceeding the threshold established in published Alzheimer's disease biomarker studies (measured by nanoneedle biosensor or equivalent immunoassay).
* We will also establish the cut off values of pTau217 of plasma based on the data from 20 AD patients and 30 normal control participants.

  * Time Frame: At single sample collection

Secondary Outcome Measures:

* Ratio of pTau217 to total Tau across plasma samples
* Distribution of pTau217 levels in the donor population

Biospecimen Retention:

Samples will be analyzed for biomarker levels; aliquots may be stored for future biomarker validation studies.

Eligibility Criteria:

* Inclusion: De-identified human plasma samples from standard blood bank donations
* Exclusion: Samples failing quality control or insufficient volume

Study Population:

Approximately 250 de-identified donated plasma samples obtained from healthy adult blood donors.

Estimated Enrollment: 250 samples

ELIGIBILITY:
Inclusion Criteria:

* The plasma sample from donators.

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Anybody who can donate blood.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Tau and pTau | 6 months.
  Concentration of Tau and pTau217 in plasma.
Concentration of pTau217 and Tau | 6 months.
  We will use nanoneedle technology to measure the concentration of Tau and pTau217 in collected plasma samples from blood donators.

CONTACTS AND LOCATIONS:
Overall Officials: Zhongcong Xie, M.D., Ph.D., Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
We do not know the names of any blood donators who provide samples of plasma.

REFERENCES:
- [Result] 40. Tatebe H, Kasai T, Ohmichi T, et al. Quantification of plasma phosphorylated tau to use as a biomarker for brain Alzheimer pathology: pilot case-control studies including patients with Alzheimer's disease and down syndrome. Mol Neurodegener. Sep 4 2017;12(1):63. doi:10.1186/s13024-017-0206-8 41. Mielke MM, Hagen CE, Xu J, et al. Plasma phospho-tau181 increases with Alzheimer's disease clinical severity and is associated with tau- and amyloid-positron emission tomography. Alzheimers Dement. Aug 2018;14(8):989-997. doi:10.1016/j.jalz.2018.02.013 42. Janelidze S, Mattsson N, Palmqvist S, et al. Plasma P-tau181 in Alzheimer's disease: relationship to other biomarkers, differential diagnosis, neuropathology and longitudinal progression to Alzheimer's dementia. Nat Med. Mar 2020;26(3):379-386. doi:10.1038/s41591-020-0755-1 43. Karikari TK, Pascoal TA, Ashton NJ, et al. Blood phosphorylated tau 181 as a biomarker for Alzheimer's disease: a diagnostic performance and prediction modelling study using data from four prospective cohorts. Lancet Neurol. May 2020;19(5):422-433. doi:10.1016/S1474-4422(20)30071-5 44. Palmqvist S, Insel PS, Stomrud E, et al. Cerebrospinal fluid and plasma biomarker trajectories with increasing amyloid deposition in Alzheimer's disease. EMBO Mol Med. Dec 2019;11(12):e11170. doi:10.15252/emmm.201911170 45. Palmqvist S, Janelidze S, Quiroz YT, et al. Discriminative Accuracy of Plasma Phospho-tau217 for Alzheimer Disease vs Other Neurodegenerative Disorders. JAMA. Aug 25 2020;324(8):772-781. doi:10.1001/jama.2020.12134 46. Janelidze S, Berron D, Smith R, et al. Associations of Plasma Phospho-Tau217 Levels With Tau Positron Emission Tomography in Early Alzheimer Disease. JAMA Neurol. Nov 9 2020;doi:10.1001/jamaneurol.2020.4201 47. Thijssen EH, La Joie R, Strom A, et al. Plasma phosphorylated tau 217 and phosphorylated tau 181 as biomarkers in Alzheimer's disease and frontotemporal lobar degeneration: a retrospective diagnostic performance study. Lan